CLINICAL TRIAL: NCT03383965
Title: A Clinical Study of CD30 Targeted CAR-T in Treating CD30-Expressing Lymphomas
Brief Title: CD30 Targeted CAR-T in Treating CD30-Expressing Lymphomas
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Immune Cell, Inc. (Industry)
Collaborators: Weifang People's Hospital (Other)
Responsible Party: Principal Investigator, Xiulian Sun, Principal Investigator, Immune Cell, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD30-targeting CAR-T
Record Dates: First submitted 2017-12-06; First posted 2017-12-27 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-03

CONDITIONS: Hodgkin Lymphoma; Anaplastic Large Cell Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic | interventions — Biological Products

STUDY DESIGN:
Masking Description: None (Open Label)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICAR30 T cells (Experimental): anti-CD30 CAR-T cells. Patients receive ICAR30 T cells infusion.
  Interventions: Biological: ICAR30 T cells

INTERVENTIONS:
Biological: ICAR30 T cells — T cells were isolated from peripheral blood from patients enrolled. T cells were transduced with lentivirus bearing anti-CD30 antibody scFV and the activation signals of second generation CART designation. The CART cells were infused into the patients by IV with an escalating dosage.
  Other Names: Biological drug

SUMMARY:
CAR-T cells have been validated effective in treating CD19 positive B cell lymphoma. Other lymphomas like Hodgkin's lymphoma and anaplastic large cell lymphoma are CD30 positive. In this study, a newly CD30 targeted CART therapy ICAR30 is designed to specifically kill those CD30 expressing malignancies including Hodgkin's lymphoma and CD30+ anaplastic large cell lymphoma. The subjects will receive several doses of autologous ICAR30 T cells infusion and then the safety, treating effects and lasting period of these cells in vivo will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Hodgkin's lymphoma, anaplastic large cell lymphoma and other CD30 positive malignancies, relapsed or refractory:

* Karnofsky or Lansky score >50;
* Expected survival>12 weeks;
* Hgb > 8.0;
* FEV1, FVC and DLCO ≥50% of expected corrected for hemoglobin;
* LVEF≥50%;
* Creatinine<2.5mg/dl;
* Bilirubin<2.5mg/dl;
* ALT (alanine aminotransferase)/AST (aspartate aminotransferase)<3 fold normal;
* Patients must sign an informed consent.

Exclusion Criteria:

* Pregnant or lactating;
* Uncontrolled active infection including hepatitis B or C;
* HIV positive;
* Active clinically significant CNS dysfunction;
* Current use of systemic steroids;
* Heterogenous lymphocyte treatments within recent 6 months;

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Measure the safety of ICAR30 T cells | 2 years
  To assess the adverse events of ICAR30 T cells infusion in patients with Hodgkin's lymphoma and CD30+ anaplastic large cell lymphoma.

SECONDARY OUTCOMES:
Measure the anti-tumor effect of ICAR30 T cells | 3 years
  To assess the anti-tumor effect of ICAR30 T cells infusion in patients with Hodgkin's lymphoma and CD30+ anaplastic large cell lymphoma.
Measure the survival time of ICAR30 T cells in vivo | 5 years
  To measure the survival time of ICAR30 T cells in vivo, extra blood will be drawn from patients receive ICAR30 T cells infusion in the follow-up time.

CONTACTS AND LOCATIONS:
Locations (1):
- Weifang People's Hospital, Weifang, Shandong, China

IPD SHARING:
Plan to Share IPD: No